CLINICAL TRIAL: NCT01360229
Title: Acupuncture as a Symptomatic Treatment for Fatigue in Parkinson's Disease
Brief Title: Acupuncture for Fatigue in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-0533
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-07

CONDITIONS: Parkinsons Disease
Keywords: Parkinsons Disease; Fatigue
MeSH Terms: conditions — Parkinson Disease; Fatigue | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Randomized Subjects receive a sham acupuncture. (Sham Comparator): Subjects will be randomized in a 1:1 ratio to receive either real or sham acupuncture.
  Interventions: Other: Acupuncture to treat fatigue in Parkinson disease
- Randomized Subjects receive real acupuncture. (Active Comparator): Subjects will be randomized in a 1:1 ratio to receive either real or sham acupuncture.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Subjects will be randomized in a 1:1 ratio to receive real acupuncture. Acupuncture is a procedure in which specific body areas are pierced with fine needles for therapeutic purposes
  Arms: Randomized Subjects receive real acupuncture.
Other: Acupuncture to treat fatigue in Parkinson disease — Subjects will be randomized in a 1:1 ratio to receive sham acupuncture.
  Arms: Randomized Subjects receive a sham acupuncture.

SUMMARY:
This is a single-center, double-blind, placebo-controlled trial to see if acupuncture can safety and effectively treat fatigue in Parkinson's Disease (PD). Eligible subjects will receive either real or sham acupuncture twice weekly for six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PD
* Patients 40-99 years of age
* Patients who have significant fatigue
* Patients must be on a stable medication regimen for the treatment of PD

Exclusion Criteria:

* Patients who have had previous acupuncture within the past six months
* Patients who have had deep brain stimulation (DBS)
* Patients with dementia, depression, or sleep disorder
* Patients who are currently taking medications known to affect fatigue, such as stimulants

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2010-08; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benzi Kluger, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- See also: Related Info — http://www.michaeljfox.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomized Subjects Receive Real Acupuncture.: Subjects will be randomized in a 1:1 ratio to receive either real or sham acupuncture.
  Acupuncture: Subjects will be randomized in a 1:1 ratio to receive real acupuncture.
  Acupuncture is a procedure in which specific body areas are pierced with fine needles for therapeutic purposes
Period: Overall Study
Arm/Group | Randomized Subjects Receive a Sham Acupuncture. | Randomized Subjects Receive Real Acupuncture.
Started | 47 | 47
Completed | 44 | 45
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Randomized Subjects Receive a Sham Acupuncture.: Subjects were randomized in a 1:1 ratio to receive either real or sham acupuncture.
  Acupuncture to treat fatigue in Parkinson disease: Subjects will be randomized in a 1:1 ratio to receive sham acupuncture.
- Randomized Subjects Receive Real Acupuncture.: Subjects were randomized in a 1:1 ratio to receive either real or sham acupuncture.
  Acupuncture: Subjects will be randomized in a 1:1 ratio to receive real acupuncture.
  Acupuncture is a procedure in which specific body areas are pierced with fine needles for therapeutic purposes
- Total: Total of all reporting groups
Arm/Group | Randomized Subjects Receive a Sham Acupuncture. | Randomized Subjects Receive Real Acupuncture. | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (13.0) | 64.4 (10.3) | 63.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 29 | 30 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 47 | 47 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 47 | 47 | 94
Region of Enrollment [Number; unit: count of participants]
  United States | 47 | 47 | 94
Modified Fatigue Impact Scale Total [Mean (Standard Deviation); unit: units on a scale] — The range of the score is 0-84 with higher scores reflecting more severe fatigue.
  units on a scale | 50.0 (12.9) | 48.7 (10.5) | 49.4 (11.7)
Unified Parkinson Disease Rating Scale (UPDRS)-Motor subscale [Mean (Standard Deviation); unit: units on a scale] — The range of the score is 0-108 with higher scores reflecting more severe motor dysfunction due to Parkinson's disease.
  units on a scale | 26.7 (11.1) | 21.6 (7.8) | 24.2 (10.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Modified Fatigue Impact Scale Total (MFIS) Between Treatment Groups
Description: The primary outcome measure will be the change between the baseline visit and 6-week time point in the Modified Fatigue Impact Scale Total (MFIS) between treatment groups. The range of the score is 0-84 with higher scores reflecting more severe fatigue.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Randomized Subjects Receive a Sham Acupuncture. | Randomized Subjects Receive Real Acupuncture.
Number analyzed (Participants) | 47 | 47
units on a scale | -13.2 (13.8) | -16.0 (15.1)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Randomized Subjects Receive a Sham Acupuncture. | Randomized Subjects Receive Real Acupuncture.
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 1/47 | 0/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Randomized Subjects Receive a Sham Acupuncture. (N=47) | Randomized Subjects Receive Real Acupuncture. (N=47)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) — temporary increase in constipation, resolved with cessation of acupuncture

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No